CLINICAL TRIAL: NCT00227201
Title: The Association Between the Use of Complementary and Alternative Medicine and Medication Adherence in Hypertensive African-Americans
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 0301005948
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension
Keywords: African-American; Hypertension; Complementary medicine; Medication adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

INTERVENTIONS:
Behavioral: Self-affirmation intervention

SUMMARY:
The objective of this study is to better understand strategies used by African Americans with hypertension in order to control their blood pressure.

DETAILED DESCRIPTION:
The objective of this study is to better understand strategies used by African Americans with hypertension in order to control their blood pressure. Through the use of qualitative interviews, the beliefs and attitudes toward complementary medicine of African Americans with hypertension will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be African-American adults 18 years or older who were diagnosed with poorly controlled hypertension as defined by the 6th Joint National Committee guidelines (systolic >140 and diastolic >90).
2. Patients will also be eligible if they are taking any prescribed anti-hypertensive medications.
3. Patients must be able to provide informed consent in English. Participants will be recruited from Cornell Internal Medicine Associates, the primary care and general medicine practice at Cornell Medical Center, the same site as the parent grant.

Exclusion Criteria:

1. Patients who refused to participate.
2. Patients who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-06; Study Completion 2005-05

PRIMARY OUTCOMES:
The impact of positive affect induction and self-affirmation on medication adherence and blood pressure control.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Moore, Principal Investigator — Weill Medical College of Cornell University; Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Medical College, New York, New York, United States

REFERENCES:
- [Background] JA Moore, Factors that influenced medication adherence among African-Americans with hypertension, to be presented at the 12th Annual NHLBI Cardiovascular Minority Research Supplement Awardee Session, American Heart Association, November 2004.